CLINICAL TRIAL: NCT07398066
Title: DEXmedetomidine for Postoperative Analgesia and Delirium Prevention After NEUROsurgery: A Double-blinded Randomised Placebo-controlled Trial (DEX-NEURO Trial)
Brief Title: DEXmedetomidine for Postoperative Analgesia and Delirium Prevention After NEUROsurgery (DEX-NEURO Trial)
Acronym: DEX-NEURO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Ka Ting Ng, Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16023
Record Dates: First submitted 2026-01-26; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Neurosurgery; Brain Cancer; Meningioma
Keywords: dexmedetomidine; precedex; neurosurgery; delirium; pain
MeSH Terms: conditions — Brain Neoplasms; Meningioma; Delirium; Pain | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous dexmedetomidine (Active Comparator): Intravenous dexmedetomidine loading dose 0.5mcg/kg followed by 0.5mcg/kg/hour
  Interventions: Drug: Dexmedetomidine
- Intravenous normal saline (Placebo Comparator): intravenous normal saline loading and infusion dose
  Interventions: Drug: Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Dexmedetomidine — intravenous dexmedetomidine loading dose 0.5mcg/kg followed by 0.5mcg/kg/hour
  Other Names: Precedex
  Arms: Intravenous dexmedetomidine
Drug: Normal Saline (0.9% NaCl) — Intravenous normal saline loading and infusion dose of normal saline
  Arms: Intravenous normal saline

SUMMARY:
Post-craniotomy pain is common and often undertreated. Inadequate analgesia can lead to patient discomfort and higher opioid consumption, which may result in respiratory depression, sedation risks and impaired neurological assessment in the early postoperative period. The incidence of post-operative delirium after intracranial surgery was 19%, ranging from 12 to 26% caused by variation in clinical features and delirium assessment methods1. It is associated with increased morbidity, longer length of hospital stay, and harm to self or staffs.

Dexmedetomidine (Precedex) is a highly selective α2-adrenergic agonist with the properties of analgesia, sedative, anxiolytic and neuroprotection without significant respiratory depression. Most of the trials administered a loading dose of 0.5-1.0 μg/kg intravenous dexmedetomidine over 10 minutes followed by infusion dose 0.2-0.7 μg/kg/hour. The use of intraoperative dexmedetomidine is believed to reduce the usage of postoperative opioids where frequent neurological assessment is often required in neurosurgical patients. Beyond the benefit of analgesia, perioperative dexmedetomidine has been studied for prevention of postoperative delirium. Randomized trials in mixed noncardiac surgical populations reported that low-dose perioperative dexmedetomidine may reduce the incidence of delirium. Dexmedetomidine produces dose-dependent bradycardia and hypotension, which should be carefully monitored to maintain the cerebral perfusion pressure in brain surgery. However, most trials and meta-analyses have focused on general surgical or cardiac cohorts; the evidence remains limited in neurosurgical (craniotomy) patients.

Although it showed promising benefits of analgesia and neuroprotection in non-neurosurgical patients, recent meta-analyses of intraoperative dexmedetomidine reported high degree of heterogeneity due to the inclusion of varied procedures (elective vs emergent craniotomy), dosing regimes (loading dose only versus loading dose + infusion versus infusion only) and varied primary endpoints (postoperative pain scores, cumulative opioid consumption or incidence of delirium). Therefore, this randomized, double-blind, placebo-controlled trial is designed to examine the use of intravenous dexmedetomidine in the reduction of postoperative pain score and delirium in neurosurgical patients. We hypothesised that intravenous dexmedetomidine reduces postoperative pain score and delirium with lower need of rescue analgesia and amount of morphine consumption in patients undergoing craniotomy.

DETAILED DESCRIPTION:
There are several similar studies been conducted in the literature search. However, the majority of the studies focus on the intensive care unit patient or non-neurosurgery patients. It is believed that intravenous dexmedetomidine can reduce the postoperative pain score with lesser need for rescue analgesia and morphine consumption to facilitate postoperative neurological assessment.

ELIGIBILITY:
Inclusion Criteria:

* All adult (American Society of Anaesthesiologists (ASA 1-2) who >18 years old and <65 years old undergoing elective craniotomy

Exclusion Criteria:

* Patients who are ASA 3-5 or BMI <18/ >40 or allergic to dexmedetomidine will be excluded. Patients with high-grade heart block or uncontrolled bradyarrhythmia will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-07-22 (Estimated); Primary Completion 2027-07-22 (Estimated); Study Completion 2027-08-22 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score at recovery area | In the recovery area after pushing out from the operation theatre (Post-operative 1-hour, Day 1, Day 2)
  Numerical Rating Scale (0 no pain-10 most pain)

SECONDARY OUTCOMES:
Need of rescue analgesia | In the recovery area after pushing out from operation theatre (Post-operative 1-hour)
  Need to receive additional analgesia (bolus of ketamine, fentanyl, morphine) in the recovery area
Total usage of postoperative morphine use in the first 24-hour | In the first 24-hour after surgery in neurointensive care unit
  The amount of morphine usage in milligram
Postoperative nausea or vomiting | Within the first 24-hour in neurointensive care unit
  Incidence of nausea or vomiting in the first 24-hour in neurointensive care unit
Incidence of delirium | Day-1 and Day-2 in neurointensive care unit
  Assessed by CAM-ICU scoring test
Patient satisfaction scale of analgesia control | Day-1 in neurointensive care unit
  Numerical rating scale (0 not satisfy - 10 very satisfy)
Adverse events of dexmedetomidine (hypotension and bradycardia). | During surgery when intravenous dexmedetomidine is started
  systolic blood pressure < 90, heart rate <60

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Su X, Meng ZT, Wu XH et al. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery : a randomised , double-blind , placebo-controlled trial. The Lancet 2016;388:1893-902
- [Background] Zhao LH, Shi ZH, Chen GQ, et al. Use of Dexmedetomidine for Prophylactic Analgesia and Sedation in Patients With Delayed Extubation After Craniotomy: A Randomized Controlled Trial. J Neurosurg Anesthesiol 2017;29:132-9
- [Background] Bielka K, Kuchyn L, Babych V, Martycshenko K, Innozemtsev O. Dexmedetomidine infusion as an analgesic adjuvant during laparoscopic сholecystectomy : a randomized controlled study. BMC Anesthesiology 2018;18:1-6
- [Background] Li X, Yang J, Nie XL et al. Impact of dexmedetomidine on the incidence of delirium in elderly patients after cardiac surgery : A randomized controlled trial. PLoS ONE 2017;12:1-15.